CLINICAL TRIAL: NCT03863327
Title: EKG Criteria and Identification of Acute Coronary Occlusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Other Study IDs: 1173733-2
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome; STEMI; STEMI - ST Elevation Myocardial Infarction; Acute Coronary Artery Thrombosis (Diagnosis); NSTEMI - Non-ST Segment Elevation MI; Non-ST Elevation Myocardial Infarction; Non ST Segment Elevation Myocardial Infarction; Non ST Segment Elevation Acute Coronary Syndrome; Non-ST Elevation Myocardial Infarction (nSTEMI); Non STEMI
Keywords: Acute Coronary Occlusion; ACO; Occlusive Myocardial Infarction; OMI; Non-occlusive Myocardial Infarction; NOMI
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Disease; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Coronary Occlusion or near-occlusion (TIMI 0-1): a. Acute occlusion proven on angiogram (an acute culprit lesion with TIMI 0-1 flow, or description of acute total thrombotic occlusion) b. Acute culprit lesion (any TIMI score) with Peak cTNI > 10 ng/mL or cTnT > 1.0 ng/mL c. If no catheterization performed (contraindicated, not compatible with goals of care, etc), then highly elevated troponin as above plus a new/presumed new focal wall motion abnormality on echocardiography d. Positive ECG findings (by any criteria) with death occurring before attempted emergent coronary angiography and autopsy confirming ACO. For cases with positive ECG findings and death before cath but NO autopsy, these will be marked and saved in a separate group, not to be used in the primary analysis.
  Interventions: Other: No intervention
- Acute Coronary Occlusion or near-occlusion (TIMI 0-2): a. Acute occlusion proven on angiogram (an acute culprit lesion with TIMI 0-2 flow, or description of acute total thrombotic occlusion) b. Acute culprit lesion (any TIMI score) with Peak cTNI > 10 ng/mL or cTnT > 1.0 ng/mL c. If no catheterization performed (contraindicated, not compatible with goals of care, etc), then highly elevated troponin as above plus a new/presumed new focal wall motion abnormality on echocardiography d. Positive ECG findings (by any criteria) with death occurring before attempted emergent coronary angiography and autopsy confirming ACO. For cases with positive ECG findings and death before cath but NO autopsy, these will be marked and saved in a separate group, not to be used in the primary analysis.
  Interventions: Other: No intervention
- Acute severe 3-vessel disease or critical left main stenosis: 1. Severe 3-vessel disease: >/=75% stenosis in all three major coronary vessels (or equivalents in the case of anatomic variants or preexisting bypass) with an acute culprit lesion (TIMI<3) or
  2. Left main stenosis > 50% (see Smith review paper for reference): acute left main culprit of any TIMI score, or any lesion of the left main with TIMI<3 or
  3. Any other cardiac catheterization findings prompting initiation of emergent coronary artery bypass grafting within the next 120 hours
  Interventions: Other: No intervention
- No evidence of acute coronary occlusion: 1. At least three sequential negative cardiac biomarkers within 24 hours of presentation
  2. cardiac catheterization showing no culprit lesion.
  3. Angiogram showing an acute culprit lesion but both no occlusion (TIMI 2 or greater) and troponins not exceeding the cutoff above
  4. If positive troponin values present but no angiography, then the patient must have echocardiography showing no wall motion abnormality and troponin values less than the above cutoff
  5. If the patient has insufficient data to classify into one of these categories, the patient must be excluded from the study as they cannot be classified as ACO or non-ACO. For example, patients with extremely high troponin but no culprit seen on cath may have acute occlusion with complete autolysis of thrombus, myocarditis, spasm, etc. Thus the investigators cannot classify them as NO ACO when the possibility of ACO remains and cannot be disproven.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There will be no intervention as a part of this protocol.

SUMMARY:
The objective of this research study is to test the accuracy of preexisting criteria versus expert interpretation for the diagnosis of acute coronary occlusion (major heart attack due to a completely blocked blood vessel). If our hypothesis proves to be true, this would provide a significant improvement in the care for patients who present to the hospital with possible symptoms of coronary ischemia (symptoms due to lack of blood flow to the heart).

The primary analysis will be designed as a multi-center, retrospective case-control study.

DETAILED DESCRIPTION:
In this retrospective, 2-center, case-control study the investigators will investigate and compare the accuracy of various ECG criteria and expert interpretation to diagnose Acute Coronary Occlusion (ACO), with an emphasis on the diagnosis of patients with ACO but without obvious ST segment Elevation Myocardial Infarction (STEMI) criteria. The investigators will use two cohorts of patients who present with symptoms consistent with acute MI, one subsequently proven to have ACO and one proven to not have ACO.

The groups will be identified by chart reviewers who will use all clinical data except the ECGs to determine, in retrospect, and using strict criteria, if the patient had ACO at the time of the ECGs to be evaluated, or not. These reviewers will be blinded to all ECGs. The diagnosis of ACO will be dependent upon angiographic occlusion. Because in many cases of ACO, the artery spontaneously opens by the time of the angiogram, the investigators will need to have surrogate endpoints: this will be culprit on the angiogram PLUS a very elevated peak troponin, as peak troponin I > 10.0 ng/mL and peak troponin T > 1.0 ng/mL are highly correlated with ACO.

The investigators will find cases of subtle STEMI (ACO without STEMI criteria) by searching for all myocardial infarction cases that underwent angiography and percutaneous coronary intervention (PCI). The investigators will attempt by various criteria to determine from all available sources other than the ECG (angiography, echo, troponins) whether the involved artery was occluded at the time of the most diagnostic ECG that was recorded while the patient had symptoms and before the angiogram. Reviewers determining ACO or not ACO will be blinded to the ECGs. The investigators will use each pre-angiogram ECG, in sequence, for analysis, to determine if expert interpretation can not only identify occlusion that is not identified by STEMI criteria, but also to find if expert interpretation can identify occlusion on an earlier ECG. Expert ECG interpreters will interpret the ECG for evidence of ACO. Their accuracy will be compared to traditional STEMI criteria and other methods of interpretation if available.

The investigators will use as controls patients with any ST elevation, or ST depression, of any etiology that are proven to NOT have occlusion. The investigators will establish absence of occlusion by a combination of objective data points including angiogram (if performed), troponins, echocardiograms, clinical course, etc. Details of the methods are below, including specific outcome definitions used to claim the presence or absence of ACO.

ELIGIBILITY:
Inclusion Criteria:

* Recorded EKG prior to cardiac catheterization

Exclusion Criteria:

* Absence of documented EKG prior to cardiac catheterization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators plan to review and include all individuals that underwent urgent or emergent cardiac catheterization over the course of one year (January 1, 2017 - December 31, 2017).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The difference in time to diagnosis of acute coronary occlusion (ACO) between the current standard of care and advanced human ECG interpretation in patients with confirmed occlusive myocardial infarction without ST elevation myocardial infarction | 1 year
  How long does it take for an expert human ECG interpreter to diagnose ACO compared to the standard of care utilizing STEMI criteria

SECONDARY OUTCOMES:
The difference in sensitivity among the occlusive myocardial infarction (OMI) cohort for experts versus ST elevation myocardial infarction (STEMI) criteria | 1 year
  The difference in sensitivity among the occlusive myocardial infarction cohort for experts versus STEMI criteria
The difference in sensitivity among the occlusive myocardial infarction (OMI) cohort for experts versus ST elevation myocardial infarction (STEMI) criteria in all studied patients | 1 year
  The difference in sensitivity among the occlusive myocardial infarction (OMI) cohort for experts versus ST elevation myocardial infarction (STEMI) criteria in all studied patients
The difference in sensitivity among the occlusive myocardial infarction (OMI) cohort for experts versus ST elevation myocardial infarction (STEMI) criteria in patients with widened QRS | 1 year
  The difference in sensitivity among the occlusive myocardial infarction (OMI) cohort for experts versus ST elevation myocardial infarction (STEMI) criteria in patients with widened QRS

OTHER OUTCOMES:
Expert accuracy (sens/spec) for acute triple vessel / left main disease acute coronary syndrome (ACS) as evidenced by global depressions with aVR elevations, other ECG changes. | 1 year
  Expert accuracy (sens/spec) for acute triple vessel / left main disease acute coronary syndrome (ACS) as evidenced by global depressions with aVR elevations, other ECG changes. Currently, there are no ECG diagnostic criteria for these entities.
Time difference in the subtle OMI group stratified based on the presence or absence of opioid pain medications. | 1 year
  Time difference in the subtle OMI group stratified based on the presence or absence of opioid pain medications.
The rate of patients with ECGs that meet STEMI criteria that then experience a delay despite positive EKG | 1 year
  The rate of patients with ECGs that meet STEMI criteria that then experience a delay despite positive EKG
Explore the rate of false positive cath lab activations | 1 year
  Explore the rate of false positive cath lab activations
Explore the rationale for correct expert ECG interpretation of OMI without STEMI criteria | 1 year
  Explore the rationale for correct expert ECG interpretation of OMI without STEMI criteria
Explore the rationale for correct expert ECG interpretation of false positive STEMI criteria | 1 year
  Explore the rationale for correct expert ECG interpretation of false positive STEMI criteria
Time from initial ECG with subtle OMI without STEMI criteria to development of ECG meeting STEMI criteria. | 1 year
  Time from initial ECG with subtle OMI without STEMI criteria to development of ECG meeting STEMI criteria.
Determine the rate of correct expert ECG interpretation of OMI without STEMI criteria | 1 year
  Determine the rate of correct expert ECG interpretation of OMI without STEMI criteria
Determine the rate of correct expert ECG interpretation of false positive STEMI criteria | 1 year
  Determine the rate of correct expert ECG interpretation of false positive STEMI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W Smith, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis
Locations (2):
- United States (2):
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Stony Brook University Hospital, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dawkins K, Busk M, Sorensen J, Mortensen LS, Maynard C, Stinnett SS, Wagner GS, Andersen HR; DANAMI-2 investigators. Association between ST segment Resolution following Fibrinolytic therapy or Intracoronary stenting, and Reinfarction in the same myocardial region in the DANAMI-2 study population. Cardiovasc Revasc Med. 2011 Mar-Apr;12(2):75-81. doi: 10.1016/j.carrev.2010.04.003. Epub 2010 Oct 20. PMID 21421184
- [Result] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Result] Jaffe AS. Third universal definition of myocardial infarction. Clin Biochem. 2013 Jan;46(1-2):1-4. doi: 10.1016/j.clinbiochem.2012.10.036. Epub 2012 Nov 2. No abstract available. PMID 23127386
- [Result] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. J Am Coll Cardiol. 2007 Nov 27;50(22):2173-95. doi: 10.1016/j.jacc.2007.09.011. No abstract available. PMID 18036459
- [Result] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686